CLINICAL TRIAL: NCT01591915
Title: A Randomized Controlled Mindfulness Based Stress Reduction Intervention in Women With Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Principal Investigator, Elisabeth Kenne Sarenmalm, Researcher, Skaraborg Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 499-09
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer, Mindfulness Based Stress Reduction, RCT, mood, cooping, health related quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MBSR self care program including weekly sessions (Experimental): Participants will participate in an 8 week course of MBSR practice of homework assignments consisting of 20 minutes sessions, 6 days/week. Participants will partake in a structured group-formatted 8 week course that patients attend once a week for an average of 2 hours.
  Interventions: Other: MBSR
- MBSR self care program (Experimental): Participants will participate in an 8 week course of MBSR practice of homework assignments consisting of 20 minutes sessions, 6 days/week.
  Interventions: Other: MBSR
- Standard care (No Intervention)

INTERVENTIONS:
Other: MBSR — Participants in Intervention 1 and Intervention 2 will participate in an 8 week course of MBSR practice of homework assignments consisting of 20 min sessions, 6 days/week. Participants will be provided information material including a book of 20 pages introduction to mindfulness training, self-instructing CD, diary and training program. Only participants in Intervention 1 will partake in a structured group-formatted 8 week course that patients attend once a week for an average of 2 h. Led by a certified MBSR instructor, these weekly group sessions are focused on participant's experiences of mindfulness, and include yoga and meditation training. Four registered nurses, skilled in patient learning, have been educated as certified MBSR instructors.
  Arms: MBSR self care program; MBSR self care program including weekly sessions

SUMMARY:
The purpose of this study is to evaluate the effect of mindfulness based stress reduction intervention in women with breast cancer

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with breast cancer after completion of adjuvant chemotherapy or radiation therapy, with/or without endocrine therapy

Exclusion Criteria:

* patients with advanced illness at diagnosis
* patients previously used MBSR

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Mindfulness Based Stress Reduction on mood disorders | up to 5 years follow up

SECONDARY OUTCOMES:
Coping capacity and health-related quality of life | up to 5 years follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Skaraborg Hospital, Skövde, Western Region, Sweden

REFERENCES:
- [Derived] Kenne Sarenmalm E, Martensson LB, Holmberg SB, Andersson BA, Oden A, Bergh I. Mindfulness based stress reduction study design of a longitudinal randomized controlled complementary intervention in women with breast cancer. BMC Complement Altern Med. 2013 Oct 2;13:248. doi: 10.1186/1472-6882-13-248. PMID 24088535